CLINICAL TRIAL: NCT06798077
Title: Chronic Airway Disease and Multimorbidity (CAM) Cohort: Protocol of a Prospective Multicenter Observational Cohort Study
Brief Title: Chronic Airway Disease and Multimorbidity Cohort
Acronym: CAM Cohort
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); First Hospital of China Medical University (Other); Henan Provincial People's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Sichuan University (Other); Southern Medical University, China (Other); Ruijin Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ting YANG, Professor, China-Japan Friendship Hospital
Other Study IDs: 2023ZD0506003
Record Dates: First submitted 2025-01-02; First posted 2025-01-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma; Bronchiectasis
Keywords: multimorbidity; COPD; asthma; bronchiectasis; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- COPD group
- Asthma Group
- Bronchiectasis Group

SUMMARY:
Background: Chronic airway diseases (CAD), including chronic obstructive pulmonary disease (COPD), asthma and bronchiectasis, are highly prevalent and cause serious disease burden. Multimorbidity is recognized to influence treatment decision and prognosis of patients with stable CAD. The impact of multimorbidity on exacerbation CAD is under investigated.

Methods: The Chronic Airway Disease and Multimorbidity (CAM) cohort study is a prospective, multicenter, observational study aiming to recruit a minimum of 2000 patients hospitalized for exacerbation of COPD, asthma or bronchiectasis. Comprehensive data, including demographics, medical history, comorbidities, lung function, echocardiography, microbiological profiles, radiology, quality of life and treatment will be collected at baseline during the hospitalization. Follow-up data indicating the impact of both CAD and multimorbidity will be collected at 1-, 3-, 6-, 9- and 12-months after hospital discharge. Biospecimens, including blood and bronchoalveolar lavage fluid, will be collected and analyzed for biomarker detecting. Primary outcome are length of hospital stay and re-exacerbation during fellow-up. Secondary outcomes include comorbidity pattern and its impact on respiratory symptoms burden, quality of life, pulmonary function and chest imaging as well as cost and healthcare utilization.

Conclusions: The knowledge generated from CAM cohort study will fill crucial gaps in understanding how multimorbidity affects CAD and facilitate evidence-based clinical practice in the future.

DETAILED DESCRIPTION:
The Chronic Airway Disease and Multimorbidity (CAM) Cohort is a nationwide, prospective, multicenter, longitudinal observational study aimed at understanding the epidemiology and impact of multimorbidity on patients hospitalized due to exacerbation of chronic airway diseases (CAD), including chronic obstructive pulmonary disease (COPD), asthma, and bronchiectasis. The study will enroll 2,000 patients across 9 medical centers in China, following their health trajectory for one year post-hospitalization.

Objective The primary objective is to assess how multimorbidity influences treatment outcomes, hospitalization length, and readmission rates in CAD patients. Secondary goals include analyzing comorbidity patterns, their effects on symptom burden, quality of life, pulmonary function, healthcare costs, and utilization.

Study Design Participants meeting inclusion criteria will be recruited through hospital advertisements and professional referrals. Upon providing informed consent, demographic, clinical, and laboratory data will be recorded during baseline hospitalization. The study employs standardized questionnaires and clinical tools such as mMRC, CAT, and SGRQ for quality-of-life assessments. Specimens, including blood, bronchoalveolar lavage fluid (BALF), and sputum, will be collected and stored for biomarker analysis. Imaging studies such as chest CT and echocardiography will evaluate disease severity and cardiac function.

Patients will be systematically followed at 1, 3, 6, 9, and 12 months post-discharge to record disease progression, treatment adherence, exacerbations, and outcomes.

Data Collection Demographics and Risk Factors: Age, gender, smoking history, family history, and occupational exposures.

Symptoms: Disease-specific tools such as CAT/mMRC(COPD), ACQ-7 (asthma) and BEST (bronchiectasis) will quantify symptom severity.

Quality of Life (QoL): SGRQ for COPD, QoL-Bronchiectasis for bronchiectasis, and mini-AQLQ for asthma patients.

Laboratory Data: Arterial blood gas, blood count, liver and renal function, inflammatory markers, and allergy panels.

Muti-morbidities: Systematic documentation of pulmonary and extrapulmonary comorbidities, including their diagnosis, treatment, and severity.

Outcome Measures: The primary outcomes are hospital length of stay and re-exacerbation rates. Secondary outcomes include changes in pulmonary function, QoL, mental health indices, imaging findings, and healthcare resource utilization.

Quality Control Data will be managed using an electronic data capture(EDC) system, with built-in validation to ensure accuracy. Periodic data audits and centralized training for research coordinators will enhance data integrity. Monitoring committees will address data discrepancies promptly.

Ethics and Dissemination The protocol complies with the Declaration of Helsinki and has received approval from ethics committees of all participating centers. The findings will inform clinical guidelines, emphasizing the integration of multi-morbidity management in CAD care.

This study bridges significant knowledge gaps in CAD management, particularly concerning multimorbidity in hospitalized patients, aiming to enhance evidence-based clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic obstructive pulmonary disease ≥40 years of age; patients with asthma and bronchiectasis ≥18 years of age;
* The primary diagnosis on admission was "acute exacerbation of chronic obstructive pulmonary disease, uncontrolled asthma, or acute exacerbation of bronchiectasis".

Exclusion Criteria:

* Patients were unable to undergo spirometry during the stabilization period;
* Expected survival is less than 1 month;
* Refusal to sign an informed consent form;
* Chest imaging showed emerging patchy infiltrating shadows, lobar or segmental solid shadows, ground glass shadows, or interstitial changes with or without pleural effusion;
* Patients with cystic fibrosis or with interstitial lung disease or other lung diseases with tractional branchial dilatation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CAM cohort study focuses on hospitalized patients with chronic airway diseases (CAD), including chronic obstructive pulmonary disease (COPD), asthma, and bronchiectasis, during acute exacerbation episodes. Participants are recruited from 9 medical centers across China, representing diverse geographic and clinical settings.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From the date of admission until discharge or death, assessed over an estimated period of 3 to 30 days.
  The length of time participants remain hospitalized from the date of admission to the date of discharge or death, whichever comes first.

SECONDARY OUTCOMES:
Acute exacerbation during follow-up | From the date of discharge to 12 months post-discharge.
  Exacerbations will be defined based on clinical criteria specific to each disease: increased respiratory symptoms requiring additional treatment.
  Measurement Tools: The number of disease exacerbation.
All cause mortality | In-hospital and from enrollment to 12 months.
  All cause mortality.
Quality of Life in COPD Patients | From enrollment to 12 months.
  Assessing quality of life in patients with COPD using validated tools. Measurement Tools: St. George's Respiratory Questionnaire (SGRQ), scores range from 0 to 100, with higher scores indicating worse quality of life.
Quality of Life in Asthma Patients | From enrollment to 12 months
  Assessing quality of life in patients with asthma using validated tools. Measurement tool: Mini Asthma Quality of Life Questionnaire (Mini-AQLQ), each question is scored from 1 to 7, with 15 questions and a total score of 105. The higher the score, the better the quality of life.
Quality of Life in Bronchiectasis Patients | From enrollment to 12 months.
  Assessing quality of life in patients with bronchiectasis using validated tools.
  Measurement tool: Bronchiectasis Health Questionnaire (BHQ), each question is scored from 1 to 7, with 10 questions and a total score of 70. The higher the score, the better the quality of life.
Lung Function | From enrollment to 12 months
  Assessment of lung function (FEV 1) over time.
Healthcare Costs | In-hospital and from enrollment to 12 months.
  Evaluation of total healthcare costs related to the treatment of CAD, including direct costs such as hospitalisation, medication and outpatient costs.
  Measurement Unit: Total cost in local currency (e.g., RMB).
Adherence to Prescribed Medications and Treatments | From enrollment to 12 months.
  Evaluation of participants' adherence to prescribed medication regimens and treatments, using patient-reported adherence and prescription records.
  Measurement Unit: Percentage of adherence (e.g., percentage of days covered).
Polypharmacy Patterns | From enrollment to 12 months.
  Analysis of the prevalence and patterns of polypharmacy, defined as the use of 2 or more medications concurrently.
  Measurement Unit: Number of concurrent medications.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, MD, Principal Investigator — China-Japan Friendship Hospital, National Center for Respiratory Medicine
Locations (9):
- China (9):
  - National Center for Respiratory Medicine, China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
The CAM cohort study has determined that individual participant data (IPD) will not be directly shared. Instead, supporting information and aggregated results will be made available in specific formats to ensure transparency while protecting participant privacy.